CLINICAL TRIAL: NCT07315776
Title: Effects of Electrical Muscle Stimulation on Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Suranaree University of Technology (Other)
Responsible Party: Principal Investigator, SEEKAOW CHURPROONG, Principal Investigator, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EP 22 081; 4961-6056 (Other: U. of Bath Biomedical Science Research Ethics Committee)
Record Dates: First submitted 2025-11-27; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Myofascial Pain Syndrome (MPS)
Keywords: Electrical Muscle Stimulation; Myofascial pain syndrome; trigger point pressure release; electromyography; pain intensity; pressure pain threshold; ultrasound images
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain | interventions — Muscle Stretching Exercises; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Treatments were administered in a computer-generated randomised order, concealed from participants.The principal researcher collected all anonymous data for blinded analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Therapist-assisted Passive stretching (PS) (Active Comparator): Passive Stretching with Therapist Assistance: The protocol consisted of three sets of stretching. Each set was performed for 10 seconds and followed by a 10-second break, totaling one minute for the single session.
  Interventions: Other: Therapist-assisted Passive stretching (PS)
- The two-combination of EMS+AS (Experimental): Electrical Muscle Stimulation (EMS) combined with Active Stretching (AS) was applied to the upper or middle trapezius muscle to facilitate muscle elongation. The protocol consisted of three sets of performing. Each set was performed for 10 seconds and followed by a 10-second break, totaling one minute for the single session.
  Interventions: Other: The two-combination of EMS+AS
- Trigger point pressure release (TPR) (Active Comparator): Trigger Point Pressure Release (TPR): TPR was directly applied to the MTP of upper or middle trapezius muscle.The protocol consisted of three sets of performing. Each set was performed for 10 seconds and followed by a 10-second break, totaling one minute for the single session.
  Interventions: Other: Trigger point pressure release (TPR)
- Trigger point pressure release combined with active stretching (TPR+AS) (Other): Trigger Point Pressure Release (TPR) combined with Active Stretching (AS) was performed either by using neck deviation for the upper trapezius muscle or by using scapula protraction for the middle trapezius muscle during TPR. The protocol consisted of three sets of performing. Each set was performed for 10 seconds and followed by a 10-second break, totaling one minute for the single session.
  Interventions: Other: Trigger point pressure release combined with active stretching (TPR+AS)
- The triple combination therapy of EMS+AS+TPR (Experimental): This triple combination therapy was applied to enhance MTP release in the upper or middle trapezius muscles. The protocol consisted of three sets of performing. Each set was performed for 10 seconds and followed by a 10-second break, totaling one minute for the single session.
  Interventions: Other: The triple combination therapy of EMS+AS+TPR
- Transcutaneous electrical nerve stimulation (TENS) (Active Comparator): Transcutaneous Electrical Nerve Stimulation (TENS) was applied on the upper or middle trapezius muscles without stretching. The protocol consisted of three sets of operating. Each set was performed for 10 seconds and followed by a 10-second break, totaling one minute for the single session.
  Interventions: Other: Transcutaneous electrical nerve stimulation (TENS)
- Sham stimulation combined with active stretching (SS+AS) (Sham Comparator): SS+AS consisted only of active stretching of the upper or middle trapezius muscle, with no electrical current applied from EMS device. Self-stretching was performed for three sets, with each 10-second stretch followed by a 10-second break, resulting in a total session time of one minute.
  Interventions: Other: Sham stimulation combined with active stretching (SS+AS)

INTERVENTIONS:
Other: Therapist-assisted Passive stretching (PS) — The therapist stretched the upper trapezius muscle via shoulder depression and neck deviation. The middle trapezius muscle was stretched using scapular protraction while simultaneously stabilizing the mid-spine and gently pulling the arm inward.
  Other Names: PS
  Arms: Therapist-assisted Passive stretching (PS)
Other: The two-combination of EMS+AS — Electrical Muscle Stimulation combined with Active Stretching: The EMS component utilized parameters of 20 Hz frequency and 100 µs pulse width, with the amplitude adjusted individually for intensity. The EMS electrodes were placed across the muscle fibers with a 1 cm inter-electrode distance. This placement was specifically designed to restrict the electrical field, thereby inducing a local muscle contraction that opposes the direction of the active stretch being performed concurrently.
  Other Names: EMS+AS
  Arms: The two-combination of EMS+AS
Other: Trigger point pressure release (TPR) — Trigger point Pressure Release (TPR): The therapist utilized a PAIN TEST™ FPX series pressure gauge (Wagner Instruments). A round rubber 1 cm2 force gauge probe was applied directly on the MTP by gradually increasing the pressure until the participant reached their maximum pressure tolerance level.
  Other Names: TPR
  Arms: Trigger point pressure release (TPR)
Other: Trigger point pressure release combined with active stretching (TPR+AS) — Trigger point Pressure Release combined with Active Stretching (TPR+AS) was performed by applying active stretching of the trapezius muscle concurrently with TPR, using the same protocol as the standalone TPR intervention.
  Other Names: TPR+AS
  Arms: Trigger point pressure release combined with active stretching (TPR+AS)
Other: The triple combination therapy of EMS+AS+TPR — Electrical Muscle Stimulation combined with Active Stretching during Trigger point Pressure Release (EMS+AS+TPR): This triple combination therapy utilized the EMS+AS component protocol concurrently with the TPR intervention, applying the identical protocols established for the standalone EMS+AS and TPR procedures.
  Other Names: EMS+AS+TPR
  Arms: The triple combination therapy of EMS+AS+TPR
Other: Transcutaneous electrical nerve stimulation (TENS) — Transcutaneous Electrical Nerve Stimulation (TENS) was applied using the conventional protocol (60 Hz,100 µs,5 mA) with two electrodes placed directly over the MTP region, without stretching.
  Other Names: TENS
  Arms: Transcutaneous electrical nerve stimulation (TENS)
Other: Sham stimulation combined with active stretching (SS+AS) — Sham stimulation combined with active stretching (SS+AS): Participants performed AS using the same EMS device and electrode placement as in the EMS+AS protocol. However, no electrical current was applied. The procedure began with a conversation about the treatment from the researcher while the current amplitude was reduced from 1 mA to 0 mA during the trapezius muscle stretching, accompanied by a beeping sound to simulate stimulation. Participants were subsequently informed that this was the intended treatment.
  Other Names: SS+AS
  Arms: Sham stimulation combined with active stretching (SS+AS)

SUMMARY:
The goal of this clinical trial is to determine if Electrical Muscle Stimulation (EMS) combined with Active Stretching (AS) (EMS+AS) and EMS+AS combined with Trigger Point Pressure Release (TPR) (EMS+AS+TPR) are effective treatments for Myofascial Pain Syndrome (MPS) in working adults. The study will also assess the safety of the EMS+AS intervention. The main questions it aims to answer are: Do EMS+AS and EMS+AS+TPR lead to greater pain reduction, increased pressure pain threshold, and improved surface electromyography (sEMG) activity when compared to standard treatments? Furthermore, what is the participant feedback regarding EMS+AS and other treatments?

Researchers will compare EMS+AS to passive stretching (PS) and TPR to see if EMS+AS and EMS+AS+TPR are effective in treating myofascial trigger points in the trapezius muscle.

Participants will receive seven interventions across a single visit, including PS, EMS+AS, TPR, TPR combined with AS (TPR+AS), EMS+AS+TPR, Sham stimulation, and Transcutaneous Electrical Nerve Stimulation (TENS). Each treatment will consist of three 10-second sets with a 10-second rest between sets, and a 2-minute break provided between different treatments. Participants will have measurements taken on changes in pain intensity, pressure pain threshold, and sEMG activity during trapezius action pre- and post-treatment. Additionally, participants will report personal information, previous MPS treatments, and baseline health status, and provide feedback on satisfaction, treatment preferences, exercise knowledge for MPS prevention, and qualitative comments. For supplementary data, we selected only the EMS+AS and TPR interventions with the same protocol to evaluate changes in range of motion and changes in trigger point size and trapezius thickness (both at rest and during stretching) via ultrasound imaging.

DETAILED DESCRIPTION:
The main study measures included changes in pain intensity, pressure pain threshold, and sEMG activity. The supplementary study measures included ultrasound images and range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years old with either active or latent myofascial trigger points in the trapezius muscle were diagnosed with MPS by a General Practitioner (GP).
* Participants have no history of chronic diseases (cancer, cervical nerve root compression, heart arrhythmias, including hyperthyroid, muscle weakness, seizure, skin infection at the upper back, spinal cord injury, stroke).
* Participants have ability to move the upper limbs.
* Participants reported no use of pacemakers or strong pain relievers, no allergies to metals, gels, or cleaning products, and no pre-existing severe muscle soreness.

Exclusion Criteria:

* Participants less 18 years old with no myofascial trigger points in the trapezius muscle.
* Participants to have history of chronic diseases (cancer, cervical nerve root compression, heart arrhythmias, including hyperthyroid, muscle weakness, seizure, skin infection at the upper back, spinal cord injury, stroke).
* Participants cannot move the upper limbs.
* Participants reported use of pacemakers or strong pain relievers, and allergies to metals, gels, or cleaning products, and pre-existing severe muscle soreness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Changes in Pain intensity | Baseline and Day 1 (immediately post-intervention)
  Changes in pain intensity before and after treatment were measured using a numeric rating scale (0-10), where 0 represents no pain and 10 represents the worst possible pain. A reduced score indicates a better outcome.
Changes in pressure pain threshold | Baseline and Day 1 (immediately post-intervention)
  Changes in pressure pain threshold between before and after treatment were measured using a digital algometer (Wagner, Greenwich, USA). Pressure pain threshold was measured in kilogram force (kgf) or kilograms per square centimeter (kg/cm²). An increased score indicates a better outcome.
Changes in median frequency of EMG activity | Baseline and Day 1 (immediately post-intervention)
  Changes in the median frequency of surface electromyography (EMG) before and after treatment were recorded in hertz (Hz) using a 16-channel sEMG (Delsys Trigno Maize Sensor system). Changes in median frequency reflect physiological changes in muscle function. An increase in median frequency during trapezius muscle activity indicates physiological improvement.
% maximum volunatary contraction (MVC) improvement | Baseline and Day 1 (immediately post-intervention)
  %MVC improvement of EMG activity before and after treatment was recorded in percent (%) after calculating the root mean square normalized to pre-treatment values using a 16-channel sEMG (Delsys Trigno Maize Sensor system). An increase in %MVC during trapezius muscle activity indicates muscle function improvement.

SECONDARY OUTCOMES:
Changes in range of motion (ROM) of neck deviation | Baseline and Day 1 (immediately post-intervention)
  Changes in ROM of neck deviation before and after treatment were assessed through photographic analysis. Photographs of participants are analyzed using ImageJ software, and ROM was recorded in degrees. An increase in ROM indicates improved upper trapezius muscle flexibility.
Changes in myofascial trigger point (MTP) size | Baseline and Day 1 (immediately post-intervention)
  Changes in MTP size before and after treatment were assessed via ultrasound imaging and analyzed using ImageJ software. MTP size was recorded in square millimeters (mm²). A decrease in MTP size indicates improved treatment outcomes.
Changes in echointensiy at the myofascial trigger point (MTP) | Baseline and Day 1 (immediately post-intervention)
  Changes in echo intensity at the MTP before and after treatment were assessed via ultrasound imaging and analyzed using ImageJ software. The echo intensity at the MTP was recorded in pixels. Changes in echo intensity reflect transient alterations in fluid accumulation or tissue structure due to fibrotic remodeling at the MTP. An increase in MTP echo intensity indicates decreased fluid accumulation, which may predict an improved treatment outcome.
Changes in trapezius muscle thickness | Baseline and Day 1 (immediately post-intervention)
  Changes in trapezius muscle thickness at rest and during stretching were assessed via ultrasound imaging and analyzed using ImageJ software. Trapezius muscle thickness was recorded in millimetre. The observed reduction in TM thickness at rest and during stretching suggests decreased muscle tension, reflecting muscle tone improvement following treatment.

OTHER OUTCOMES:
Particpants' feedback | Day 1 (Post-treatment assessment)
  Feedback questionnaires were administered to assess participant satisfaction, treatment preferences, exercise knowledge for MPS prevention, and qualitative comments. The qualitative data derived from the participants' feedback were organized into three structural domains-overall impression, lack of satisfaction, and suggestions for improvement-which emerge directly from a careful review and categorization of recurring themes within the participants' verbatim comments.

CONTACTS AND LOCATIONS:
Overall Officials: SEEKAOW CHURPROONG, MD., Principal Investigator — University of Bath, United Kingdom.
Locations (1):
- Department of Electronic and Electrical Engineering, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No
"Participants' data being shared within the research team", as noted in the consent form. Data will not be shared with other researchers unless they formally join the research team.

REFERENCES:
- See also: Main Study Protocol — https://drive.google.com/file/d/1T_dydVByLSEM3fn5ycD5gBfc-VaC6iuS/view?usp=sharing
- See also: Main Study Ethics Amendment — https://drive.google.com/file/d/1d_zp0P5UHoa_wIXfzEcOM8Eyf6jBoFSL/view?usp=sharing
- See also: Ultrasound Study Protocol — https://drive.google.com/file/d/18X-V6BgkTwPWQqteMW_dpMvY8rpyAcJj/view?usp=sharing
- See also: Ultrasound Study Ethics Letter (Supplementary Data) — https://drive.google.com/file/d/1hurWgeXyuiyEmkWHXMUXOg7D_JpMgY6e/view?usp=sharing